CLINICAL TRIAL: NCT05908305
Title: Study of Tramadol Addiction Impact on Dental Anesthesia Succes.
Brief Title: Impact of Tramadol Addiction On Dental Anesthesia Success
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Algiers (Other)
Responsible Party: Principal Investigator, Mohammed Amir Rais, Principal Investigator, University of Algiers
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Tramadol Addict Impact On Dent
Record Dates: First submitted 2022-12-04; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Dental Pain and Sensation Disorder; Anesthesia, Local; Addiction, Opioid
Keywords: Tramadol; Addiction; Local Anesthesia; Dentistry; Carpule
MeSH Terms: conditions — Toothache; Sensation Disorders; Opioid-Related Disorders; Behavior, Addictive | interventions — Carticaine; Epinephrine; Anesthesia, Dental; Mepivacaine

STUDY DESIGN:
Intervention Model Description: Assessing local dental anesthesia success while performing different dental care among Algerian males addicted or not addicted to tramadol.
Who Masked: Care Provider
Masking Description: Dentists providing dental care participating in the study are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tramadol Addicted Patients (Active Comparator): It represents the group of tramadol addicted patients seeking dental care that require dental anesthesia.
  Interventions: Drug: articaine@ (4% 1:100000 epinephrine) dental anesthesia
- Non addicted patients (Active Comparator): The group of patients requiring dental care with local anesthesia and who are not addicted to tramadol.
  Interventions: Drug: articaine@ (4% 1:100000 epinephrine) dental anesthesia

INTERVENTIONS:
Drug: articaine@ (4% 1:100000 epinephrine) dental anesthesia — Administration, calculation and adjustment of dental local anesthesia doses.
  Other Names: mepivacaine@ (2%@ 1:100000 epinephrine) dental anesthesia

SUMMARY:
The aim is to investigate and to find a correlation between tramadol addiction misuse among Algerian males and Dental Local Anesthesia success while performing dental care and oral surgeries.

DETAILED DESCRIPTION:
Local anesthesia is by far the most important part of pain control in dentistry, it is the cornerstone that makes many dental procedures possible, not only for the patient but also for the dentist and dental hygienists. Since the pain and the dentist are almost synonymous for the patient, this makes dental anesthesia the most widely administered drugs in the dental clinics. Hence, the failure of local anesthesia in oral medicine presents an undesirable outcome both for the patient and for the practitioner.

The intraoperative pain being prevented by the administration of a local anesthesia must be followed by the management of the postoperative pain which can be often intense and thus requiring drugs administration. These drugs could be nonopioid or opioid analgesics which are also frequently used in general medicine as Tramadol.

Tramadol is 2-(dimethyl amino)-methyl)-1-(3'-methoxyphenyl) cyclohexanol hydrochloride. It is 4-phenyl-piperidine analogue of the opioid drug codeine. It is generally well tolerated with few and rare side effects. Moreover, comparative studies have mostly shown that Tramadol is more effective than NSAIDs for post operative pain control. However, its misuse is increasingly growing and has become obvious in Algeria.

Tramadol addiction has become very frequent, and its unjustified use is expanding. This might be attributed to the fragility of the health system and the replacement of the qualified pharmacists by non-qualified helpers or assistants.

ELIGIBILITY:
Inclusion Criteria:

* Males
* ≥18 years old <65
* Without comorbid conditions (Hypertension, diabetes, Asthma etc..)
* Tramadol addicted (regular tramadol user)
* Only tramadol addicted, if any other drugs are regularly consumed, the patient is excluded.

Exclusion Criteria:

* Females
* ˂ 18 years old
* With comorbid conditions (HTN, diabetes, epilepsy etc..)
* ≥ 65 years old men.
* Not addicted to tramadol or addicted to other drugs with it.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males will be recruited since this topic is somehow stigma in Algeria. Drugs abusive use in Algeria is found among males and females but considered for religious and society related reasons a stigma.
Enrollment: 300 (Estimated)
Dates: Start 2023-06-10 (Estimated); Primary Completion 2023-09-29 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Measuring in (ML) the quantity of dental anesthesia used in each participants group to achieve analgesic effect | 3 months
  The quantity (ml) of dental anesthesia used to perform dental and oral surgery procedure among tramadol addicted and non-addicted patients will be mesured to investigate the difference.
To determine the number of dental anesthesia carpules used for each group participants during dental and oral procedures | 3 months
  Among addicted and non-addicted patients, the number of carpules of dental anesthesia necessary for total analgesic effect will be determined.

SECONDARY OUTCOMES:
To determine the quantity ( mg) of tramadol and the time of consumption ( in months) necessary to cause dental anesthesia failure among addicted patients. | 3 months
  As our hypothesis suggested that tramadol addiction cause dental anesthesia failure, we would like to calculate the dose and number of months of tramadol consumption necessary to provok dental anesthesia failure as an addiction complication

REFERENCES:
- [Background] Carnaval TG, Sampaio RM, Lanfredi CB, Borsatti MA, Adde CA. Effects of opioids on local anesthesia in the rat: a codeine and tramadol study. Braz Oral Res. 2013 Nov-Dec;27(6):455-62. doi: 10.1590/S1806-83242013000600003. PMID 24346042
- [Background] Guven M, Mert T, Gunay I. Effects of tramadol on nerve action potentials in rat: comparisons with benzocaine and lidocaine. Int J Neurosci. 2005 Mar;115(3):339-49. doi: 10.1080/00207450590520948. PMID 15804720
- [Background] Premnath S, Alalshaikh G, Alfotawi R, Philip M. The Association Between Coffee Consumption and Local Anesthesia Failure: Social Beliefs and Scientific Evidence. Cureus. 2020 Apr 24;12(4):e7820. doi: 10.7759/cureus.7820. PMID 32467795
- [Background] Fung EY, Giannini PJ. Implications of drug dependence on dental patient management. Gen Dent. 2010 May-Jun;58(3):236-41; quiz 242-3. PMID 20478804